CLINICAL TRIAL: NCT00069966
Title: A Phase II Trial of BBR 2778 in Combination With Cytarabine, Methylprednisolone and Cisplatin (BSHAP) as Salvage in Patients With Relapsed Aggressive Non-Hodgkin's Lymphoma
Brief Title: Pixantrone, Cytarabine, Methylprednisolone, and Cisplatin in Treating Patients With Aggressive Non-Hodgkin's Lymphoma in First Relapse
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316466; THERADEX-AZA-II-02; CWRU-NOVU-1403; SUNY-HSC-4849; NOVUSPHARMA-AZA-II-02
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2004-11

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; anaplastic large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Burkitt Lymphoma | interventions — Filgrastim; Rituximab; Cisplatin; Cytarabine; Methylprednisolone; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: cisplatin
Drug: cytarabine
Drug: methylprednisolone
Drug: pixantrone dimaleate
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pixantrone, cytarabine, methylprednisolone, and cisplatin, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have relapsed aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of pixantrone, cytarabine, methylprednisolone, and cisplatin in patients with aggressive non-Hodgkin's lymphoma in first relapse.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the validity and safety of this regimen as a mobilization regimen before high-dose chemotherapy with stem cell support in these patients.

OUTLINE: This is an open-label, multicenter study.

* Salvage therapy: Patients receive pixantrone IV over 1 hour on day 1; cisplatin IV over 30 minutes on days 1-4; methylprednisolone IV over 15-30 minutes on days 1-5; and cytarabine IV over 2 hours on day 5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After 2 courses of salvage therapy, patients are re-evaluated and treated as follows:

* Complete response (CR) or partial response (PR): Patients with a CR or PR who are suitable candidates for autologous stem cell transplantation (ASCT) proceed to mobilization therapy, high-dose chemotherapy, and ASCT. Patients with a CR or PR who are unsuitable candidates for ASCT continue to receive salvage therapy for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Stable disease: Patients with stable disease continue to receive salvage therapy for up to 6 courses. Patients who have a CR or PR after 3-4 courses of salvage therapy and who are suitable candidates for ASCT proceed to mobilization therapy, high-dose chemotherapy, and ASCT off study at the investigator's discretion.

  * Mobilization therapy (optional regimen; regimen used for mobilization is at the investigator's discretion): Patients receive rituximab* IV on days 1 and 7; pixantrone IV over 1 hour on day 2; cisplatin IV over 30 minutes on days 2-5; cytarabine IV over 2 hours on day 6; and methylprednisolone IV over 15-30 minutes on days 2-6. Patients also receive filgrastim (G-CSF) subcutaneously once daily beginning on day 7 and continuing until blood counts recover. Patients receive 1 or more courses of mobilization therapy during which stem cells are harvested. Patients then proceed to high-dose chemotherapy and subsequent re-infusion of harvested stem cells.

NOTE: *If this mobilization regimen is used, patients with T-cell lymphoma do not receive rituximab

* High-dose chemotherapy and ASCT: Patients receive high-dose chemotherapy and ASCT per institutional standard practice.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma (NHL)

  * Any stage, with or without B symptoms
  * The following subtypes are eligible:

    * Diffuse large cell (B and T cell types)
    * Anaplastic large cell
    * Diffuse mixed cell
    * Immunoblastic large cell
    * Follicular large cell
    * Transformed follicular NHL
    * Diffuse aggressive not otherwise classified
    * Burkitt-like lymphoma
* Bone marrow positive or negative
* At least 1 measurable lesion

  * Patients with bone marrow as the only site of disease are eligible without a measurable lesion
* No more than 1 episode of progressive disease, occurring after a response (complete response [CR], complete response unconfirmed [CR_u], or partial response [PR]) to prior chemotherapy* NOTE: *Patients with less than a CR, CRu, or PR and no progression, but who are good candidates for high-dose chemotherapy with stem cell support may be eligible (will be decided on an individual basis)
* No chemotherapy-refractory disease, defined as follows:

  * Stable or progressive disease documented at restaging immediately after the completion of induction therapy
* No lymphoblastic lymphoma, or mantle cell lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3* NOTE: *Lower values may be accepted if clearly due to bone marrow involvement by lymphoma

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)*
* AST or ALT no greater than 2.0 times ULN*
* Alkaline phosphatase no greater than 2.0 times ULN*
* No history or clinical symptoms of hepatitis B or hepatitis C virus

  * Patients with seropositivity due to prior vaccination for hepatitis B are eligible NOTE: *Higher values may be accepted if clearly due to liver involvement by lymphoma

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* LVEF at least 50% by MUGA
* No clinically significant cardiovascular abnormalities
* No New York Heart Association grade II-IV cardiovascular disease
* No myocardial infarction within the past 6 months
* No severe cardiac arrhythmia
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* HIV negative
* No clinically significant neurological abnormalities
* No condition that would preclude study safety or interfere with study results
* No concurrent serious uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior rituximab immediately after the first chemotherapy regimen allowed

Chemotherapy

* See Disease Characteristics
* See Biologic therapy
* At least 6 months since prior anthracycline therapy (e.g., cyclophosphamide, doxorubicin, vincristine, and prednisone [CHOP])
* More than 2 years since prior fludarabine
* More than 2 years since prior nitrosoureas
* More than 1 year since prior platinum-based chemotherapy or cytarabine, unless a CR or CR_u was achieved
* No prior cumulative dose of cisplatin greater than 600 mg/m^2
* No prior single or cumulative dose of doxorubicin greater than 450 mg/m^2

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the whole pelvis
* No prior radioimmunotherapy

Surgery

* More than 4 weeks since prior major thoracic and/or abdominal surgery
* At least 1 week since prior minor surgery

Other

* Recovered from prior therapy

  * Alopecia allowed
  * Grade 1 peripheral neuropathy allowed
* More than 30 days since prior participation in another investigational drug study
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Vose, MD, Study Chair — University of Nebraska
Locations (29):
- United States (28):
  - Arizona Oncology Associates - Craycroft Road Offices, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Rocky Mountain Cancer Centers - Colorado Springs, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Delaware Clinical & Laboratory Physicians, Newark, Delaware
  - Pasco, Hernando Oncology Associates, P.A., New Port Richey, Florida
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Piedmont Hematology-Oncology Associates, Winston-Salem, North Carolina
  - Gabrail Cancer Center - Canton Office, Canton, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cancer Care Associates-West, Oklahoma City, Oklahoma
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fairfax Northern Virginia Hematology Oncology, P.C. - Fairfax, Fairfax, Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Hospital Auxilio Mutuo, Hato Rey, Puerto Rico